CLINICAL TRIAL: NCT04849468
Title: Effect of Preemptive Intramuscular Diclofenac on Minimal Effective-Dose Bupivacaine Saddle Block for Minor Perianal Surgeries
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Hitham Mohammed Aly Elsayed, Anesthesia consultant, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2019-01-187-KFUH
Record Dates: First submitted 2021-04-08; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: patients will be randomly allocated into two groups; Diclofenac (D) group which will receive 75 mg (3ml) IM Diclofenac in a 5ml syringe and Saline (S) group which will receive 3ml IM saline in a similar 5ml syringe
Who Masked: Participant, Outcomes Assessor
Masking Description: The studied drugs will be prepared immediately before injection by an anesthesiologist blinded to the study methodology and will be administered by a second blinded anesthesiologist patients and assessor also will be unaware of the type of group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diclofenac (D) group (Active Comparator): Diclofenac (D) group which will receive 75 mg (3ml) intramuscular Diclofenac in a 5ml syringe in the holding area 30 minutes before spinal block
  Interventions: Drug: Declofenac
- Saline (S) group (Active Comparator): Saline (S) group which will receive 3ml intramuscular saline in a similar 5ml syringe in the holding area 30 minutes before spinal block
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Declofenac — evaluating the preemptive effect of intramuscular declofenac on postoperative analgesia in patients undergoing perianal surgeries under saddle block
  Arms: Diclofenac (D) group
Drug: saline — evaluating the preemptive effect of intramuscular saline on postoperative analgesia in patients undergoing perianal surgeries under saddle block as control
  Arms: Saline (S) group

SUMMARY:
The research will be carried out in order to test the effect of Intramuscular (IM) Diclofenac, administered as preemptive analgesic with minimal effective dose spinal anesthesia in perianal surgeries, on prolonging the time to first request for analgesic and lowering analgesic consumption. Investigators hypothesized that using IM Diclofenac in this surgery will postpone the time to first analgesic request and will decrease the consumption of post-operative analgesics. Our method includes dividing the patients into control and study groups and recording the first analgesic request and post-operative analgesic consumption after surgery and comparing the results.

DETAILED DESCRIPTION:
Effective control of post-operative pain is an issue that has been repeatedly emphasized and has received an increasing amount of attention in the past few years (1, 2). Opioids, despite their side effects, are still the main cornerstone in managing acute postoperative pain (3). Preemptive analgesia refers to the administration of effective analgesia prior to surgical trauma. The main mechanism of preemptive analgesia is desensitization of the central nervous system and prevention of pain before its onset. (3). Non-opioid preemptive analgesics are commonly used to increase analgesic efficacy and patient satisfaction as well as to reduce opioid consumption and side effects. Saddle anesthesia is a selective spinal anesthesia that is commonly used for perianal surgeries (4-7).

Investigators previously performed a prospective up-down sequential allocation study to evaluate the minimum effective dose of hyperbaric bupivacaine that is needed for inducing a satisfactory and reliable saddle block for perianal surgeries that was restricted to the most caudal spinal nerve roots (S4-coccygeal) that supply the perianal region (8). Although the block produced no motor block in the lower limbs (thus allowing early ambulation), rapid sensory recovery resulted in early request of analgesia and increased opioid consumption. In this prospective, randomized, double blinded, placebo controlled clinical trial, Investigators hypothesize that a single dose of IM diclofenac administered before spinal anesthesia, will decrease postoperative pain, and delay and reduce postoperative analgesic requirement in patients undergoing minor perianal surgeries under minimal effective-dose bupivacaine saddle block

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I and II scheduled for elective outpatient perianal surgery in the lithotomy position (hemorrhoidectomy, fistulectomy)

Exclusion Criteria:

* contraindications to regional anesthesia, bleeding disorders, are morbidly obese, suffer from mental health problems, are on analgesic medication or psychotropic drugs, have a known history of allergy to amide local anesthetic drugs, if there is a language barrier, or if they are unwilling to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | up to 24 hours
  visual analogue scale
Time to first analgesia request | up to 24 hours
  first request of analgesia by the patient
total consumption of analgesia | 24 hours
  total consumption of tramadol in mg

CONTACTS AND LOCATIONS:
Locations (1):
- King Fahd University Hospital, Khobar, Eastern Province, Saudi Arabia